CLINICAL TRIAL: NCT00410852
Title: Randomized Study to Evaluate the Efficacy and Safety of Two Endovenous Insulin Protocols and a Subcutaneous Insulin Protocol in Critically Ill Patients
Brief Title: Efficacy and Safety of Three Insulin Protocols in Medical Intensive Care Unit Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAPESP 2005/50557-5
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Intensive Care
Keywords: Insulin; Hyperglycemia; Hypoglycemia; Intensive care; Critical care
MeSH Terms: conditions — Insulin Resistance; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Procedure: Computer-assisted IV insulin infusion protocol (algorithm A)
- B (Experimental)
  Interventions: Procedure: Leuven Strict glycemic control protocol (Algorithm B)
- C (Active Comparator)
  Interventions: Procedure: Conventional Intermittent Insulin Protocol (Algorithm C)

INTERVENTIONS:
Procedure: Computer-assisted IV insulin infusion protocol (algorithm A) — Computer assisted insulin protocol (CAIP), with continuous intravenous insulin adjustments aiming blood glucose levels between 100 mg/dl and 130 mg/dl.
  Arms: A
Procedure: Leuven Strict glycemic control protocol (Algorithm B) — Leuven protocol: continuous intravenous insulin infusion aimiming blood glucose levels between 80mg/dl and 110mg/dl.
  Arms: B
Procedure: Conventional Intermittent Insulin Protocol (Algorithm C) — Conventional treatment: intermitent subcutaneous insulin according to a sliding scale, starting with blood glucose levels higher than 150mg/dl.
  Arms: C

SUMMARY:
To evaluate the efficacy and safety of three insulin algorithms in medical ICU patients (MICU).

DETAILED DESCRIPTION:
Strict glycemic control has been recommended for critically ill patients. However, its implementation may face difficulties with increased nursing workload, inadequate glucose control and higher risk of hypoglycemia.

We designed a computer guided protocol to adjust endovenous insulin infusion aiming glucose levels between 100mg/dl and 130 mg/dl. This trial evaluates the efficacy and safety of this protocol (algorithm A), compared to a standard endovenous insulin infusion protocol (algorithm B) and a conventional subcutaneous insulin protocol (algorithm C).

Methods : MICU patients with at least one blood glucose ≥ 150 mg/dL and who are on mechanical ventilation, or had SIRS, or are admitted because of trauma or burn will be randomized to one of the following treatments: algorithm A - continuous insulin infusion with adjustments guided by hand held device or desktop software targeting glucose levels between 100mg/dL-130mg/dL; algorithm B - continuous insulin aiming glucose levels between 80mg/dl-110mg/dl using Van den Berghe's insulin protocol; algorithm C - conventional treatment - intermittent subcutaneous administration of insulin if blood glucose levels exceeds 150mg/dL; insulin will be administered as IV boluses in hypotensive patients.

The randomization list was generated in blocks of six by computer software. Patients will be randomly assigned in a 1:1:1 ratio to have their glucose controlled by one of the three insulin algorithms with the use of a central, computerized system accessed by Internet, permitting concealment of allocation list. Randomization will be stratified according to study site.

The study is planned to enroll 165 patients in order to have 80% power to detect a 20mg/dl difference in blood glucose means between groups, assuming standard deviation equal to 33 mg/dl and two-tailed alpha equal to 0.05. Efficacy will be measured by the mean of patients' median blood glucose and safety measured by the incidence of hypoglycemia (≤40 mg/dL). Analysis will follow the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Criteria 1, 2 and 3 must be present:

  1. Clinical patients admitted to an Intensive Care Unit
  2. At least one blood glucose measurement >= 150 mg/dL (capilar, venous or arterial blood)
  3. At least one of the following:

     1. Patient on mechanical ventilation for an acute process, with expected duration of mechanical ventilation of at least 24 hours
     2. Polytrauma patients
     3. Severe burn patients
     4. Systemic Inflammatory Response Syndrome (modified criteria), with at least three of the following: core temperature >=38°C or <=36°C; heart rate >=90 beats/min, except in patients with a medical condition or receiving a medication known to prevent tachycardia; respiratory heart rate >= 20 breaths/min or a PaCO2 <=32mmHg, or the use of mechanical ventilation for an acute process; white-cell count of >=12.000/mm3 or <=4.000/mm3 or a differential count showing >10% percent immature neutrophils

        Exclusion Criteria:
* Age < 21 years
* Surgical patients (surgery less than 24hs before admission to ICU)
* Diabetic ketoacidosis
* Non-ketotic hyperosmolar state
* Patients with defined diagnosis of brain death
* Moribund state in which death is perceived to be imminent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2005-05; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Efficacy: mean of patients' median blood glucose during ICU stay | ICU Stay
Safety: incidence of hypoglycemia (≤40 mg/dL)during ICU stay | ICU stay

SECONDARY OUTCOMES:
Death from any cause | ICU and in-hospital
ICU and hospital length of stay | ICU and in-hospital
Five-day variation in SOFA score | Five days
90-day health status | 90 days
Days on mechanical ventilation
Initiation of dialysis
Days on antibiotics
Days on inotropic of vasopressor support
Necessity of red blood cell transfusions
Bilirubin peak
Platelets through

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre B Cavalcanti, MD, Study Chair — Hospital Israelita Albert Einstein; Eliezer Silva, PhD, Study Director — Hospital Israelita Albert Einstein; Jose Eluf-Neto, PhD, Study Director — Departamento de Medicina Preventiva, Faculdade de Medicina da Universidade de Sao Paulo; Milton Caldeira, MD, Principal Investigator — Hospital Regional Sao Jose; Glauco Westphal, MD, Principal Investigator — Centro Hospitalar UNIMED
Locations (5):
- Brazil (5):
  - Complexo Hospitalar UNIMED, Joinville, Santa Catarina
  - Hospital Dona Helena, Joinville, Santa Catarina
  - Hospital Regional Sao Jose, Joinville, Santa Catarina
  - Hospital Estadual Mario Covas, Santo André, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo